CLINICAL TRIAL: NCT04145193
Title: A Phase 2, Open-label, Randomized, Multicenter, Platform Study of Novel Oncology Therapies in Combination With Adjuvant Chemotherapy in High-risk, Microsatellite-stable Colorectal Cancer (COLUMBIA-2)
Brief Title: Novel Oncology Therapies in Combination With Adjuvant Chemo in High-risk MSS-CRC
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study withdrawn prior to enrollment due to changing standard of care landscape.
Sponsor: MedImmune LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: D910CC00002
Record Dates: First submitted 2019-10-16; First posted 2019-10-30 (Actual); Last update posted 2020-09-21 (Actual); Status verified 2020-09

CONDITIONS: Microsatellite-stable Colorectal Cancer
Keywords: Microsatellite stable; Colon Cancer; colorectal cancer; MSS-CRC; adjuvant
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms | interventions — Folfox protocol; Oxaliplatin; Leucovorin; Fluorouracil; durvalumab; monalizumab

STUDY DESIGN:
Intervention Model Description: The study is designed to evaluate the efficacy and safety of standard-of-care adjuvant mFOLFOX6 chemotherapy alone or in combination with novel oncology therapies. The study will be conducted in subjects who have undergone radical surgical resection for Stage II or III MSS-CRC, are eligible for mFOLFOX6 adjuvant therapy, and are confirmed as ctDNA positive post-surgery.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Control Arm (mFOLFOX6) (Active Comparator): Parts of mFOLFOX6 are: Oxaliplatin 85 mg/m2 IV infusion Q2W (Day 1 of every 14-day cycle), Folinic acid (leucovorin) 400 mg/m2 IV infusion Q2W (Day 1 of every 14-day cycle), Fluorouracil (5-FU) 400 mg/m2 IV bolus on Day 1 then 2,400 mg/m2 over 46 to 48 hours IV infusion Q2W (Day 1-2 of every 14-day cycle).
  Interventions: Drug: Standard of Care - mFOLFOX6; Drug: E1 - mFOLFOX and durvalumab; Drug: E2 - mFOLFOX6, durvalumab and oleclumab; Drug: E3 - mFOLFOX6, durvalumab and monalizumab
- Durvalumab (Experimental): Durvalumab 1500 mg IV, Q4W (Day 1 of every other 14-day cycle)
  Interventions: Drug: E1 - mFOLFOX and durvalumab; Drug: E2 - mFOLFOX6, durvalumab and oleclumab; Drug: E3 - mFOLFOX6, durvalumab and monalizumab
- Oleclumab (Experimental): Oleclumab 3,000 mg IV Q2W x5 then Q4W (Day 1 of every 14-day cycle through cycle 4 then Day 1 of every other 14-day cycle)
  Interventions: Drug: E2 - mFOLFOX6, durvalumab and oleclumab
- Monalizumab (Experimental): Monalizumab 750 mg IV, Q2W (Day 1 of every 14-day cycle)
  Interventions: Drug: E3 - mFOLFOX6, durvalumab and monalizumab

INTERVENTIONS:
Drug: Standard of Care - mFOLFOX6 — Parts of mFOLFOX6 are: Oxaliplatin 85 mg/m2 IV infusion Q2W (Day 1 of every 14-day cycle), Folinic acid (leucovorin) 400 mg/m2 IV infusion Q2W (Day 1 of every 14-day cycle), Fluorouracil (5-FU) 400 mg/m2 IV bolus on Day 1 then 2,400 mg/m2 over 46 to 48 hours IV infusion Q2W (Day 1-2 of every 14-day cycle).
  Other Names: FOLFOX (Oxaliplatin, Folinic acid (leucovorin), Fluorouracil (5-FU))
  Arms: Control Arm (mFOLFOX6)
Drug: E1 - mFOLFOX and durvalumab — Parts of mFOLFOX6 are: Oxaliplatin 85 mg/m2 IV infusion Q2W (Day 1 of every 14-day cycle), Folinic acid (leucovorin) 400 mg/m2 IV infusion Q2W (Day 1 of every 14-day cycle), Fluorouracil (5-FU) 400 mg/m2 IV bolus on Day 1 then 2,400 mg/m2 over 46 to 48 hours IV infusion Q2W (Day 1-2 of every 14-day cycle).
  Durvalumab 1500 mg IV, Q4W (Day 1 of every other 14-day cycle)
  Other Names: Durvalumab (MEDI-4736)
  Arms: Control Arm (mFOLFOX6); Durvalumab
Drug: E2 - mFOLFOX6, durvalumab and oleclumab — Parts of mFOLFOX6 are: Oxaliplatin 85 mg/m2 IV infusion Q2W (Day 1 of every 14-day cycle), Folinic acid (leucovorin) 400 mg/m2 IV infusion Q2W (Day 1 of every 14-day cycle), Fluorouracil (5-FU) 400 mg/m2 IV bolus on Day 1 then 2,400 mg/m2 over 46 to 48 hours IV infusion Q2W (Day 1-2 of every 14-day cycle).
  Durvalumab 1500 mg IV, Q4W (Day 1 of every other 14-day cycle) Oleclumab 3,000 mg IV Q2W x5 then Q4W (Day 1 of every 14-day cycle through cycle 4 then Day 1 of every other 14-day cycle)
  Other Names: Durvalumab (MEDI-4736) + Oleclumab (MEDI-9447)
  Arms: Control Arm (mFOLFOX6); Durvalumab; Oleclumab
Drug: E3 - mFOLFOX6, durvalumab and monalizumab — Parts of mFOLFOX6 are: Oxaliplatin 85 mg/m2 IV infusion Q2W (Day 1 of every 14-day cycle), Folinic acid (leucovorin) 400 mg/m2 IV infusion Q2W (Day 1 of every 14-day cycle), Fluorouracil (5-FU) 400 mg/m2 IV bolus on Day 1 then 2,400 mg/m2 over 46 to 48 hours IV infusion Q2W (Day 1-2 of every 14-day cycle).
  Durvalumab 1500 mg IV, Q4W (Day 1 of every other 14-day cycle) Monalizumab 750 mg IV, Q2W (Day 1 of every 14-day cycle)
  Other Names: Durvalumab (MEDI-4736) + Monalizumab (IPH2201)
  Arms: Control Arm (mFOLFOX6); Durvalumab; Monalizumab

SUMMARY:
Columbia 2 is a Phase 2 platform study to evaluate the safety and efficacy of standard of care (FOLFOX) alone and in combination with novel oncology therapies in adjuvant high-risk microsatellite-stable colorectal cancer

DETAILED DESCRIPTION:
Columbia 2 is a Phase 2, open-label, randomized, multicenter, platform study of novel oncology therapies in combination with adjuvant chemotherapy in patients with high-risk microsatellite-stable colorectal cancer.

ELIGIBILITY:
Inclusion Criteria

1. Written informed consent and any locally required authorization obtained from the subject/legal representative prior to performing any protocol-related procedures, including screening evaluations.
2. Age ≥ 18 years at the time of screening
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
4. Histologically proven Stage II or Stage III CRC

   Subjects must also meet the following criteria:
   1. Eligible for 6 months of mFOLFOX6 adjuvant chemotherapy within 8 weeks after surgery
   2. Must NOT have received prior systemic chemotherapy, immunotherapy, or radiotherapy for treatment of CRC.
   3. Must NOT have defective DNA mismatch repair (MSI) as documented by testing
5. Margin-negative (R0; defined as >1 mm clearance) surgical resection
6. Postoperative ctDNA-positive status defined by the presence of ctDNA derived from plasma; determined using a validated assay per protocol
7. Subjects must have adequate organ function
8. Body weight > 35 kg
9. Adequate method of contraception per protocol

Exclusion Criteria:

1. Any condition that, in the opinion of the investigator, would interfere with evaluation of the investigational product or interpretation of subject safety or study results.
2. Evidence of metastatic disease (including presence of tumor cells in ascites or peritoneal carcinomatosis resected "en bloc").
3. History of allogeneic organ transplantation.
4. Active or prior documented autoimmune disorders within the past 5 years as noted in the protocol.
5. Cardiac and vascular criteria:

   1. History of venous thrombosis within the past 3 months prior to the scheduled first dose of study treatment.
   2. Presence of acute coronary syndrome including myocardial infarction or unstable angina pectoris, other arterial thrombotic event including cerebrovascular accident or transient ischemic attack or stroke within the past 6 months prior to the scheduled first dose of study treatment.
   3. New York Heart Association (NYHA) Class II or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or uncontrolled hypertension.
   4. History of hypertensive crisis/hypertensive encephalopathy within the past 6 months prior to the scheduled first dose of study treatment.
   5. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥ 470 ms
6. Uncontrolled intercurrent illness, see the protocol for details.
7. History of another primary malignancy except for: (a) Malignancy treated with curative intent and with no known active disease ≥ 5 years prior to the scheduled first dose of study treatment and of low potential risk for recurrence
8. History of active primary immunodeficiency.
9. Active infection including tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus.
10. Known allergy or hypersensitivity to any of the investigational product or noninvestigational product formulations.
11. Any condition that, in the opinion of the investigator, would prevent the initiation of 6 months adjuvant therapy within 8 weeks of surgery
12. Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment.
13. Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to the scheduled first dose of study treatment, or anticipation of the need for major surgical procedure during the course of the study.
14. Current or prior use of immunosuppressive medication within 14 days prior to the scheduled first dose of study treatment.

Ages: 18 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2024-03-19 (Estimated); Study Completion 2024-03-19 (Estimated)

PRIMARY OUTCOMES:
ctDNA clearance | From the time of first dose to 6 months post treatment
  ctDNA clearance is defined as the change from ctDNA positive status at baseline to ctDNA negative post baseline (6 months)

SECONDARY OUTCOMES:
Incidence of adverse events | From time of first dose to 90 days post last dose
  The secondary endpoint of safety as assessed by the number of subjects with adverse events and serious adverse events
Disease free survival | From time of first dose till end of study (5 years)
  From randomization until time of first documented incidence of disease recurrence, secondary cancer, or death due to any cause, whichever occurs first
Disease free survival at 12 months | From time of first dose till end of study (5 years)
  Percentage of subject who are disease free at 12 months post first dose of treatment
overall survival | From time of first dose till end of study (5 years)
  From randomization until death due to any cause
Serum conenctration levels of novel agents in combination with mFOLFOX6 | From Day 1 up to 90 days post last dose
  Pharmacokinetics of novel agents in combination with FOLFOX
Number of subjects with detectable anti-drug antibody (ADA) to novel agents in combination with mFOLFOX6 | From Day 1 up to 90 days post last dose
  Immunogenicity of novel agents in combination with mFOLFOX6

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment:
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at
  https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home